CLINICAL TRIAL: NCT04873921
Title: Immediate Effects of Sterile Kinesio Tape Applied During Anterior Cruciate Ligament Reconstruction on Edema, Pain and Range of Motion
Brief Title: Effects of Sterile Kinesio Tape on Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Associated Proffesor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA 21/133
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Pain; Edema
Keywords: Kinesiotape; Anterior Cruciate Ligament Reconstruction; Edema; Pain; Range of Motion
MeSH Terms: conditions — Pain, Postoperative; Edema; Pain

STUDY DESIGN:
Intervention Model Description: Patients are randomized into 2 groups; Group 1: Sterile Kinesio tape application (n=28), Group 2: Control group (n=28). Group 1 will receive Sterile Kinesio Taping application within 72 hours applied with Sterile Web Cut Kinesio Tape without tension additional to standard postoperative care. Group 2 will receive only standard postoperative care.
Who Masked: Participant, Outcomes Assessor
Masking Description: Group 1 and 2 will be assessed and treated by two different experienced physiotherapists for each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Sterile Kinesio tape application (Experimental): Sterile Kinesio Taping application will be applied with Sterile Web Cut Kinesio Tape (Sterile Kinesio Tex Tape, Alberquerque, USA) without tension.
  Interventions: Other: sterile kinesio taping
- Group 2: Control group (No Intervention): Group 2 will not receive any taping

INTERVENTIONS:
Other: sterile kinesio taping — Application area will be cleaned and dried prior to application to increase the adhesiveness of the tape and application will be done by an experienced physiotherapist during ACLR surgery.
  Other Names: taping
  Arms: Group 1: Sterile Kinesio tape application

SUMMARY:
Anterior cruciate ligament reconstruction (ACLR) is a surgical tissue graft replacement of the anterior cruciate ligament, located in the knee, to restore its function after an injury. ACLR is used as the gold standard in coping with pain, deformity, and instability for the patients. The most important factors affecting the success of both surgery and postoperative rehabilitation programs are edema, joint movement limitation and pain around the knee in the early postoperative period. If these parameters are managed well in the postoperative period, the quality of life of the patient increases much earlier. In this respect, kinesio taping treatment, which is practical, comfortable, and safe for the patient, is one of the complementary treatment modalities with positive clinical results. No researchers have studied the effects of Sterile Kinesio Tape applied during ACL reconstruction on edema, pain and range of motion in immediate care postoperatively. The purpose of our study İS to assess effects of Sterile Kinesio Tape application on postoperative edema, pain and range of motion after ACLR within 72 hours. Thirty-seven patients who have undergone ACLR will be recruited to our study. Patients will be randomized into 2 groups; Group 1: Sterile Kinesio tape application, Group 2: Control group. All patients will be assessed for pain intensity (with Visual Analog Scale-VAS), edema (with tape measurement) and range of motion (with goniometric measurement-knee flexion/extension). Assessments will be done every day for 3 days (a total of 3 measurements). Group 1 will receive Sterile Kinesio Taping application within 72 hours applied with Sterile Web Cut Kinesio Tape without tension additional to standard during ACLR postoperative care. Group 2 will receive only standard postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent anterior cruciate ligament reconstruction

Exclusion Criteria:

* with soft tissue or bone problems affecting the hip or ankle
* who any neurologic problems,
* who had any systematic rheumatic problems,
* had scoliosis,
* who had undergone orthopedic surgery before,
* who were obese (BMI> 30 kg/m2)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 3 days
  Pain intensity will be assessed (every day for 3 days) with Visual Analog Scale (VAS). VAS is a 10-cm line with no marks along it, anchored with the words "no pain" on one hand, and "the most severe pain" on the other. Patients will be simply instructed to place a mark along the line at a level representing the intensity of their pain during activity
Edema Assessment | 3 days
  Edema will be assessed (every day for 3 days) with circumferential measurements in centimeters using basic tape measurement for ACLR knees at 5 levels: incision level, upper part of incision (5 cm above and 10 cm above) and lower part of incision (5 cm below and 10 cm below)
Range of motion measurement | 3 days
  Range of motion measurement will be done (every day for 3 days) with universal goniometry for knee flexion and extension. Knee flexion and extension movements will be measured in the supine position for both knees. The measurements will be recorded in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided